CLINICAL TRIAL: NCT00808665
Title: Does Continuous Perioperative Dexmedetomidine Infusion Reduce Time to Discharge in Patients Undergoing Major Lumbar Fusion? A Double-Blind, Placebo-Controlled Study
Brief Title: Intraoperative Infusion of Precedex to Reduce Length of Stay After Lumbar Spine Fusion
Acronym: DEXREDLOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-081331
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Results first posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Spinal Fusion Acquired; Spinal Stenosis; Lesions of Lumbosacral Intervertebral Disc; Spinal Diseases
Keywords: Lumbar Fusion; Inflammation; Dexmedetomidine; Length of Hospital Stay; General Anesthesia; Anti-inflammatory; GPCR; Cytokine; Immune Response
MeSH Terms: conditions — Spinal Stenosis; Spinal Diseases; Inflammation | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Experimental): At the beginning of spinal surgery, patients will receive 1 hour dexmedetomidine intravenous bolus of 0.7 mcg/kg, followed by infusion of dexmedetomidine at a rate of 0.5 mcg/kg/hour for 2 hours, followed by an infusion of dexmedetomidine at a rate of 0.2 mcg/kg/hour for the duration of the procedure and for 4 hours after the procedure.
  Interventions: Drug: Dexmedetomidine
- Saline (Placebo Comparator): Since this is a blinded study, at the beginning of spinal surgery, patients will receive a 1 hour 0.9% saline intravenous bolus at a rate and volume commensurate with a 0.7 mcg/kg/hour bolus of dexmedetomidine. Similarly, this will be followed with a saline infusion at a rate of 0.5 mcg/kg/hour for 2 hours, followed by an infusion of saline at a rate of 0.2 mcg/kg/hour for the duration of the procedure and for 4 hours after the procedure.
  Interventions: Drug: 0.9% Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will be given 0.7 mcg/kg/hr of dexmedetomidine over the first hour of surgery, followed by continuous infusion of 0.5 mcg/kg/hr of dexmedetomidine for the next 2 hours of surgery. Dexmedetomidine dose will be reduced to 0.2 mcg/kg/hr for the duration of the procedure and continued at that rate for four hours postoperatively. Patients in the placebo arm will receive an equal per-kg IV volume of 0.9% Sodium Chloride over the same periods. Drug administration will be controlled for both arms of the study using a continuous infusion pump.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: 0.9% Saline — Patients in the placebo arm will receive an equal per-kg IV volume of 0.9% Sodium Chloride over the same periods. Drug administration will be controlled for both arms of the study using a continuous infusion pump.
  Arms: Saline

SUMMARY:
Major lumbar spine surgery causes inflammation, soreness and swelling that can delay discharge from the hospital. Dexmedetomidine (DEX) has been shown to have anti-inflammatory effects. This study will evaluate whether DEX can help get patients out of the hospital faster after major spine surgery by reducing the inflammation associated with the procedure itself. A separate part of the study will evaluate the blood levels of some specific indicators of inflammation called cytokines. Measuring cytokines before and after surgery will aid in determining if DEX has altered the inflammatory response.

DETAILED DESCRIPTION:
Inflammation is a two-edged sword, one edge essential for healing, the other potentially delaying recovery. There is evidence that modest attenuation of the initial course of the inflammatory response (IR) - essentially "banking the fire" of the early IR - may be of benefit in shortening overall hospital course. Several medications have been evaluated/utilized intra- and perioperatively to modulate different components of IR, including local anesthetics, steroids and non-steroidal drugs. Additionally, the pro-and anti-inflammatory properties of various alpha- and beta-adrenergic agonists and antagonists have been characterized. Of this last category, dexmedetomidine (DEX), a highly specific ligand for all the subtypes of the alpha-2 receptor throughout the body, has substantial potency for sedation, analgesia and a reduction in the stress response in a wide variety of surgical environments as well as contributing to cardiovascular stability during Coronary Artery Bypass Graft (CABG) and open craniotomy. Additionally, DEX has been shown to have quite powerful anti-inflammatory activity in a murine endotoxin model. DEX's anti-inflammatory activity is likely expressed at G protein-coupled receptors (GPCRs) - either conformationally similar to, or the actual "native" alpha-2 receptor - on polymorphonuclear leukocytes, tissue macrophages, mast cells and other immune system cells. Through these receptors, DEX may attenuate the early phase of IR by limiting immune signaling or release of inflammatory cytokines, potentially favorably limiting the body's IR to injury.

In this present study, our primary assumption is that an ordinarily exuberant IR would be invoked by major spine fusion surgery. Continuous administration of intravenous DEX during and immediately after surgery might sufficiently modulate the IR to shorten hospital stay. Therefore, in a prospective, randomized, placebo-controlled, double blinded fashion, we plan to evaluate the potential for a perioperative infusion of DEX to reduce "time-to-fitness-for-discharge" (generally easier to mark and a more accurate surrogate of time-to-discharge) in patients undergoing major 3+ level lumbar spinal fusion procedures. Additionally, cytokine markers, pain scores and additional pain medication requirements associated with surgery will be measured.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Classification I - III
* Scheduled for Open Posterior Lumbar Fusion over 3+ (bony) levels

Exclusion Criteria:

* Allergy to dexmedetomidine
* Cardiac disease with reduced ejection fraction < 30%
* History of cirrhosis, active hepatitis or attenuated hepatic function
* Chronic use of steroids, COX-2 inhibitors, alpha-2 agonists, or statins
* Current anticoagulant therapy
* Patients requiring motor evoked potential (MEP) monitoring
* Positive pregnancy test

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L Blair, DO, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Taniguchi T, Kurita A, Kobayashi K, Yamamoto K, Inaba H. Dose- and time-related effects of dexmedetomidine on mortality and inflammatory responses to endotoxin-induced shock in rats. J Anesth. 2008;22(3):221-8. doi: 10.1007/s00540-008-0611-9. Epub 2008 Aug 7. PMID 18685927
- [Background] Sanders RD, Maze M. Alpha2-adrenoceptor agonists. Curr Opin Investig Drugs. 2007 Jan;8(1):25-33. PMID 17263182
- [Background] Ma D, Hossain M, Rajakumaraswamy N, Arshad M, Sanders RD, Franks NP, Maze M. Dexmedetomidine produces its neuroprotective effect via the alpha 2A-adrenoceptor subtype. Eur J Pharmacol. 2004 Oct 11;502(1-2):87-97. doi: 10.1016/j.ejphar.2004.08.044. PMID 15464093
- [Background] Nelson LE, Lu J, Guo T, Saper CB, Franks NP, Maze M. The alpha2-adrenoceptor agonist dexmedetomidine converges on an endogenous sleep-promoting pathway to exert its sedative effects. Anesthesiology. 2003 Feb;98(2):428-36. doi: 10.1097/00000542-200302000-00024. PMID 12552203
- [Background] Guo TZ, Jiang JY, Buttermann AE, Maze M. Dexmedetomidine injection into the locus ceruleus produces antinociception. Anesthesiology. 1996 Apr;84(4):873-81. doi: 10.1097/00000542-199604000-00015. PMID 8638842

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 68 participants were assessed for eligibility but 5 failed Inclusion and Exclusion criteria and were not randomized
Period: Overall Study
Arm/Group | Dexmedetomidine | Saline
Started | 31 | 32
Medication Started | 30 | 32
Completed Intra-operative Dose | 26 | 32
Completed Post Operative Doses | 25 | 29
Completed | 25 | 29
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — only required minimally invasive surgery | 1 | 0
Not completed — surgery cancelled | 1 | 0
Not completed — required an additional procedure | 0 | 1
Not completed — Physician Decision | 3 | 1
Not completed — Medication stopped by resident | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Saline | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [59 to 68] | 58 [52 to 64] | 60 [55 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 45
  Male | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  United States | 31 | 32 | 63

OUTCOME MEASURES:

1. Primary Outcome: Time Required After Surgery to Reach Fitness for Discharge From Hospital
Time Frame: Start of study drug to time to reach fitness for discharge from hospital (about 3 to 5 days)
Population: analysis done on the 54 participants that received the entire course of Dexmedetomidine or placebo.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Dexmedetomidine | Saline
Number analyzed (Participants) | 25 | 29
days | 3.2 [2.0 to 4.0] | 3.2 [2.2 to 4.6]
Statistical Analysis 1: Comparison: Dexmedetomidine vs Saline; Test type: Superiority; p = 0.36, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: from study drug start to hospital discharge ( about 3-5 days)
Description: Participants that received any amount of study drug ( "Medication Started" Milestone in participant flow) were included in Adverse Event Reporting.
Arm/Group | Dexmedetomidine | Saline
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 1/30 | 3/32
Other Adverse Events (participants affected / at risk) | 23/30 | 26/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine (N=30) | Saline (N=32)
Cardiac Arrthymia (Cardiac disorders) | 1 (1) | 1 (1)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine (N=30) | Saline (N=32)
hypotension (Cardiac disorders) | 6 (6) | 5 (5) — requiring Intravenous fluids
Bleeding (Surgical and medical procedures) | 9 (9) | 6 (6) — requiring blood transfusions
Delirium (Nervous system disorders) | 2 (2) | 1 (1)
Wound Infection (Surgical and medical procedures) | 2 (2) | 1 (1)
Return the the Operating Room (Surgical and medical procedures) | 3 (3) | 0 (0)
Device/Hardware Failure (Surgical and medical procedures) | 2 (2) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Prolonged Memory loss (Nervous system disorders) | 0 (0) | 1 (1)
EKG Changes (Cardiac disorders) | 23 (23) | 26 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes